CLINICAL TRIAL: NCT01571544
Title: The Use of Thermal Suits as Preventing Hypothermia During Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R12038
Record Dates: First submitted 2012-03-29; First posted 2012-04-05 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thermal suit (Experimental): Randomly selected half of the patients will use thermal suit prior to anesthesia, during the surgery and post anesthesia care unit.
  Interventions: Device: Thermal suit
- Conventional clothing (Active Comparator): Randomly selected half of the patients will use conventional clothing prior to anesthesia, during the surgery and post anesthesia care unit.
  Interventions: Other: Conventional clothing

INTERVENTIONS:
Device: Thermal suit — Thermal suit
  Arms: Thermal suit
Other: Conventional clothing — Conventional clothing
  Arms: Conventional clothing

SUMMARY:
Unintentional hypothermia of a patient is a common adverse effect during surgical procedures. The aim of this prospective, randomised, controlled study is to determine whether the use of thermal suit could prevent surgical patient from experiencing thermal loss than conventional measures.

Hypothesis: The investigators assume that a difference of 0.5°C in body temperature between the groups is clinically relevant.

DETAILED DESCRIPTION:
The aim of this study was to compare a thermal suit (T-Balance) and conventional warming methods to maintain a constant body temperature in patients undergoing robotic laparoscopic radical prostatectomy under general anesthesia.

A sample size calculation was made using a power analysis. Patients were randomly allocated into two groups.

Patients in the intervention group were put on the T-Balance 1 hour before anesthesia induction. Patients in the control group got conventional cotton clothes. Intra-operatively same warming methods were used in both groups. The measuring points of the temperature were esophagus (core temperature), left axilla, dorsal surface of the left middle finger and back of the left foot.

Anesthesia was induced via target-controlled infusion. All temperature data of the patients were collected and recorded electrically and continuously.

ELIGIBILITY:
Inclusion Criteria:

* radical prostatectomy, American Society of Anaesthesiologists class I-III, age 18-90

Exclusion Criteria:

* mental status with inability to give informed consent, neuromuscular disorders, Raynaud's disease, unstable angina pectoris

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Temperature | from one hour before surgery up to the ward after surgery, estimated 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sirkka-Liisa Lauronen, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland